CLINICAL TRIAL: NCT04030871
Title: A Single-Center, Investigator-Initiated, Randomized, Pilot Study Comparing Cost Effectiveness Two Commercially Available Gastric Feeding Tubes (Capsule Dome G-Tube Versus Balloon Bolus Feeding Tube).
Brief Title: A Randomized, Pilot Study Comparing Cost Effectiveness on Two Commercially Available Gastric Feeding Tubes
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Inability to recruit study participants
Sponsor: Ohio State University (Other)
Responsible Party: Principal Investigator, George Papachristou, Principal Investigator, Ohio State University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: New-41476
Record Dates: First submitted 2019-05-29; First posted 2019-07-24 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-08

CONDITIONS: Long Term Enteral Tube Feeding

STUDY DESIGN:
Intervention Model Description: A Single-Center, Investigator-Initiated, Randomized, Pilot Study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Capsule Dome G-Tube (Active Comparator): Capsule Dome G-Tube
  Interventions: Device: Capsule Dome G-Tube
- Balloon Bolus feeding tube (Active Comparator): Balloon Bolus feeding tube
  Interventions: Device: Balloon Bolus feeding tube

INTERVENTIONS:
Device: Capsule Dome G-Tube — Feeding replacement tubes with two different FDA approved devices in forty subjects
  Arms: Capsule Dome G-Tube
Device: Balloon Bolus feeding tube — Feeding replacement tubes with two different FDA approved devices in forty subjects
  Arms: Balloon Bolus feeding tube

SUMMARY:
This document is a protocol for a human research study. This study is to be conducted according to US and international standards of Good Clinical Practice (International Conference on Harmonization ICHE6, R2), the Code of Federal Regulations Title 21 parts 803 and 812, and other applicable government regulations and Institutional research policies and procedures. The purpose of the study is to compare the cost effectiveness and tolerability of standard of care gastrostomy tubes to newer capsule dome gastrostomy tubes. The newer tubes are significantly more expensive, therefore the aims of this study will be to determine economic feasibility of going to the new model. Data are lacking on the newer g-tubes in terms of longevity and cost-effectiveness

DETAILED DESCRIPTION:
Gastrostomy tubes are enteral feeding devices that are designed to provide delivery of nutrients, fluids, medications directly into the stomach, bypassing the mouth and esophagus. These devices are also known as gastrostomy tubes (G-tubes) or percutaneous endoscopic gastrostomy tube (PEG tube). These are used when patients have conditions that make them unable to swallow. While parenteral (Intravenous) nutrition and nasogastric tubes are also nutritional-support methods. A variety of g-tube designs have been used in pediatric to adult populations. The insertion of a g-tube is one of the most common endoscopic procedures and is relatively safe. The OSU endoscopy lab placed 381 g-tubes in 2018.

The most common G-tube used by the OSU Endoscopy Lab is the Balloon Bolus feeding tube. In 2017 the Capsule Dome G-Tube became commercially available. The cost of the Capsule dome g-tube is twice as expensive as the standard balloon g-tube. The insertion costs would be comparable.

The need to perform a pilot comparative study of the two g-tubes is necessary to improve our physicians understanding of the potential cost-effectiveness that longer patency we could gather from the alternative device.

ELIGIBILITY:
Inclusion Criteria:

1. Signed an IRB-approved informed consent form for the study.
2. Adults (18-75 years of age)
3. Requirement of long term enteral tube feeding (> to 12 months) and are due for a change of their initial or prior replacement bolus Percutaneous Endoscopic Gastrostomy (PEG) tube.
4. Ability to consent for the procedure and study.
5. Subjects must be able to communicate in english via telephone and understand the assessment checklists.
6. Expected to survive 12 months. Exclusion Criteria

The following subjects will not be eligible for inclusion in the study:

1. Enteral feeding is not necessary for at least 12 months,
2. A medical condition that makes it impossible for them to communicate via telephone
3. Subjects requiring feeding into the jejunum via a combined gastroenterostomy-jejunostomy tube
4. Subjects who require endoscopic replacement of their current gastrostomy tube.
5. Impaired cognition, inability to provide assessment feedback by telephone.
6. Subjects not expected to survive > 12 months

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2019-10-25 (Actual); Primary Completion 2023-12-30 (Actual); Study Completion 2023-12-30 (Actual)

PRIMARY OUTCOMES:
Comparison of PEG tube device longevity | Up to twelve months
  Time (metric is looking at Q3 month follow-up for one year)

SECONDARY OUTCOMES:
Measure the cost difference of two PEG tube devices | Up to twelve months
  Metrics evaluated using a cost-effectiveness analysis

CONTACTS AND LOCATIONS:
Overall Officials: Jeffery R Groce, MD, Principal Investigator — Ohio State University
Locations (1):
- Endoscopy Doan, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No